CLINICAL TRIAL: NCT07293234
Title: Effect of Simethicone on Helicobacter Pylori Detection: A Paired, Randomized, Pilot Study in Routine Endoscopic Practice
Brief Title: Effect of Simethicone on Helicobacter Pylori Detection in Routine Endoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, MD, DM, FJGES , Director interventional Endoscopy , senior consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SIMPACT-HP
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: H Pylori Infection
MeSH Terms: interventions — Simethicone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Simethicone Group) (Experimental)
  Interventions: Procedure: Simeticone
- Arm B (Placebo Group) (Placebo Comparator)
  Interventions: Procedure: placebo (plain water)

INTERVENTIONS:
Procedure: Simeticone — If the initial RUT (Rapid Urease Test) is positive, the patient receives 200 mL of oral simethicone (4 mg/mL). The preparation is: Each simethicone bottle contains 40 mg/mL in 10 mL volume (400 mg total per bottle). To prepare 1 litre of 4 mg/mL solution: we will take a 1 litre bottle of sterile water, aspirate and discard 100 mL, then add 10 bottles of simethicone (100 mL total volume containing 4000 mg). This creates 1000 mL of solution with a concentration of 4 mg/mL [8,9]
  After 30-60 minutes, a second endoscopy is performed and biopsies are taken for RUT, culture, PCR, and histology (Mention in detail the sites of the tissue acquisition).
  Arms: Arm A (Simethicone Group)
Procedure: placebo (plain water) — If the initial RUT is positive, the patient receives an oral placebo (200 ml water). After 30-60 minutes, a second endoscopy is performed and the same set of biopsies will be taken (pre-intervention and post-intervention biopsies)
  Arms: Arm B (Placebo Group)

SUMMARY:
Rationale: Although simethicone improves mucosal clarity, in vitro evidence suggests that its surfactant properties may disrupt bacterial adherence or viability. These findings raise concerns that simethicone may negatively affect the sensitivity of endoscopic-based H. pylori diagnostic methods. To date, no prospective in vivo study has evaluated whether simethicone influences H. pylori detection through endoscopic sampling. This randomized paired trial is designed to address this gap in evidence and evaluate whether simethicone administration reduces diagnostic yield.

Hypothesis: Simethicone administration prior to upper gastrointestinal endoscopy may reduce the detection rate of H. pylori by interfering with bacterial detection and diagnostic test performance.

Note on Pilot Study Design: This is a pilot study conducted to test feasibility and inform the design of a larger future trial.

Objectives:

To evaluate whether oral administration of simethicone prior to endoscopy reduces the diagnostic yield of H. pylori using the rapid urease test (RUT).

To evaluate whether oral administration of simethicone impacts the detection of H. pylori by other diagnostic methods, including histology, PCR, culture, and urea breath testing performed during endoscopy.

To explore variability in detection methods and determine feasibility for a future larger trial.

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years and <80 years
* Rapid Urease Test (RUT) positive on endoscopic gastric biopsy
* Ability to provide informed consent

Exclusion Criteria

* Use of antibiotics or bismuth compounds within 4 weeks prior to enrollment
* Use of proton pump inhibitors (PPIs) within 2 weeks prior to enrollment
* Use of H2 receptor blockers within 72 hours prior to enrollment
* History of previous gastric surgery
* Current anticoagulation therapy
* Severe thrombocytopenia (platelet count <50,000/mm³)
* Severe comorbidities that contraindicate the administration of sedation
* Immunodeficiency
* Pregnancy
* Negative initial Rapid Urease Test (RUT)
* Inability to provide informed consent

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in H.pylori Detection Rate by Rapid Urease Test before and After simethicone administration | Baseline ( prior to intervention ) and 30-60 minutes post- intervention (same day assessment during second endoscopy

SECONDARY OUTCOMES:
Change in H.pylori Detection Rate by Histology, PCR, Culture, and Urea Breath Test before and After Simethicone or placebo | Baseline (pre -intervention) and 30-60 minutes post- intervention
  This outcome measures the difference in detection rates of Helicobacter pylori using four additional diagnostic methods- histopathology , PCR, bacterial culture,and the urea breath test before and After administration of simethicone or placebo.The comparison will determine whether simethicone impacts these methgods similarly to RUT

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Mohan Kumar Ramchandani, MD, DM, Study Director — AIG Hospitals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bisschops R, Areia M, Coron E, Dobru D, Kaskas B, Kuvaev R, Pech O, Ragunath K, Weusten B, Familiari P, Domagk D, Valori R, Kaminski MF, Spada C, Bretthauer M, Bennett C, Senore C, Dinis-Ribeiro M, Rutter MD. Performance measures for upper gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2016 Sep;48(9):843-64. doi: 10.1055/s-0042-113128. Epub 2016 Aug 22. No abstract available. PMID 27548885
- [Result] Ahsan M, Babaei L, Gholamrezaei A, Emami MH. Simethicone for the Preparation before Esophagogastroduodenoscopy. Diagn Ther Endosc. 2011;2011:484532. doi: 10.1155/2011/484532. Epub 2011 Aug 4. PMID 21826120
- [Result] Beaufort IN, Verbeek RE, Bosman JH, Al-Toma A, Bogte A, Alvarez Herrero L, Weusten BLAM. Optimal timing of simethicone administration prior to upper endoscopy: A multicenter, single-blind, randomized controlled trial. Endosc Int Open. 2023 Oct 17;11(10):E992-E1000. doi: 10.1055/a-2157-5034. eCollection 2023 Oct. PMID 37854124